CLINICAL TRIAL: NCT02979119
Title: The European Paediatric Network for Haemophilia Management and the PedNet Haemophilia Registry
Brief Title: The European Paediatric Network for Haemophilia Management ( PedNet Registry)
Acronym: PedNet
Status: Recruiting | Type: Observational
Sponsor: PedNet Haemophilia Research Foundation (Other)
Responsible Party: Principal Investigator, Gili Kenet, Director, PedNet Haemophilia Research Foundation
Other Study IDs: Version 6.4 November 2022
Record Dates: First submitted 2014-10-21; First posted 2016-12-01 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Factor VIII Deficiency; Factor IX Deficiency
Keywords: Hemophilia; Children; Inhibitors; Prophylaxis; Long-term outcome; Congenital
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Cohort I: Children with mild ( FVIII/IX 6 to 25%), moderate (FVIII/IX 1 to 5%) or severe (FVIII/IX <1%) haemophilia A or B, born from January 1st 2000 until December 31st 2009 who have been or are to be treated with coagulation proteins in one of the participating centres
- Cohort II: Children with mild ( FVIII/IX 6 to 25%), moderate (FVIII/IX 1 to 5%) or severe (FVIII/IX <1%) haemophilia A or B, born from January 1st 2010 until December 31st 2019 who have been or are to be treated with coagulation proteins in one of the participating centres
- Cohort III: Children with mild ( FVIII/IX 6 to 25%), moderate (FVIII/IX 1 to 5%) or severe (FVIII/IX <1%) haemophilia A or B, born from January 1st 2020 until December 31st 2029 who have been or are to be treated with coagulation proteins in one of the participating centres
- Cohort IV: Cohort IV Group/Cohort Description: Children with mild ( FVIII/IX 6 to 25%), moderate (FVIII/IX 1 to 5%) or severe (FVIII/IX <1%) haemophilia A or B, born from January 1st 2030 until December 31st 2039 who have been or are to be treated with coagulation proteins in one of the participating centres

SUMMARY:
Rationale:

Haemophilia is a rare disease; to improve knowledge international collaboration is needed. Well-defined clinical data will be collected from complete cohorts in order to prevent selection bias.

Objective:

To collect data on bleeding during neonatal period, endogenous (genetic) and exogenous (treatment-related) determinants of inhibitor development and long term outcome.

DETAILED DESCRIPTION:
Design: Multicenter Prospective Observational Birth Cohort Study

Population:

Patients with haemophilia A and B with FVIII/IX levels of <1 to 25% born between 1-1-2000 and 1-1-2040.

Intervention:

No intervention; only documentation of patient characteristics and parameters of routine patient care and outcome

Main outcome parameters:

Outcome: clinically relevant inhibitor development, bleeding pattern and joint status on physical examination and imaging.

Determinants: baseline FVIII/IX levels, measurement of inhibitory antibodies, family history, FVIII/IX gene mutation, details on replacement therapy (according to each infusion for the first 50 treatment days, and annually thereafter) and surgeries.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

* No burden for the patients. Well-defined clinical data will be collected from the medical files. Participating in this registry will not change the number of visits to the clinic. All outcome parameters that are collected (including laboratory results) are part of routine clinical care.
* Direct benefit is not to be expected. However, the direct interaction between centres that treat patients with rare diseases improves both clinical care and will result in better guidelines and as such may provide indirect benefit.
* Multicentre participation: haemophilia is a very rare condition. Therefore, collecting data on a multi-centre observational cohort is the only way to study this specific population.
* The registry concerns young boys and girls with haemophilia and cannot be performed in older patients, as >90% of inhibitors occur develop during the first 50 exposure days, and the results of prophylactic replacement therapy are highly dependent on the initiation of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Haemophilia A or B
* Factor VIII/ IX activity of <1 to 25%
* Complete records of Factor treatment and bleeds
* Treated in one of the participating centres

Exclusion Criteria:

* Patients referred because of an inhibitor*
* Informed consent not obtained

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with mild ( FVIII/IX 6 to 25%), moderate (FVIII/IX 1 to 5%) or severe (FVIII/IX <1%) haemophilia A or B, born from January 1st 2000 until January 1st 2030 who have been or are to be treated in one of the participating centres
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2014-06; Primary Completion 2039-12 (Estimated); Study Completion 2039-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with antibody development to exogenous clotting factors | Until patient reaches age of 18
  Allo-antibodies against Factor VIII and IX; Blood test: measurement in Bethesda units (BU), positive according to local standards, for most labs >0.5 BU

SECONDARY OUTCOMES:
Long term outcome of haemophilia on joint status using the Hemophilia Joint Health Score (HJHS) and MRI techniques. | From diagnose every 5 years until patient reaches age of 18
  Effect of different prophylactic regimen on bleeding and joint damage
Long term outcome different Immune Tolerance Induction (ITI) therapies in patients with inhibitor. | From date first positive inhibitor titer preferably every 3 years until patient reaches age of 18
  Effect of different ITI therapies on bleeding and joint damage. Joint damage is assessed using the HJHS and MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Gili Kenet, PhD, MD, Study Director — The National Hemophilia Center Ministry of Health Sheba Medical Center Ramat Gan, Israel; Christoph Male, MD, Study Chair — Medical University of Vienna; Gili Kenet, PhD, MD, Principal Investigator — The National Hemophilia Center Ministry of Health Sheba Medical Center Ramat Gan, Israel
Locations (39):
- Austria (2):
  - Universitäts-Klinik für Kinder- und Jugendheilkunde, Graz
  - Medical University of Vienna - Department of Paediatrics, Vienna
- Service of Pediatric Haematology University Hospital Leuven, Leuven, Belgium
- Canada (2):
  - Division of Hematology/Oncology Hôpital St Justine, Montreal
  - Division of Haematology/Oncology Hospital for Sick Children, Toronto
- Czechia (2):
  - Haemophilia Comprehensive Care Centre, Centre for Thrombosis and Haemostasis Children's University Hospital Brno, Brno
  - Department of Paediatric Haematology/oncology - University Hospital Motol, Prague
- Department of Pediatrics Århus Kommunehospital Skejby Sygehus, Aarhus, Denmark
- Children's Hospital Helsinki University Hospital, Helsinki, Finland
- France (3):
  - Service Hématologique Centre Regional Traitement d'Hemophilie Bicetre, Le Kremlin-Bicêtre
  - Service d'Hématologie Pédiatrique Hôpital Universitaire La Timone, Marseille Cedex-05
  - Centre de traitement des hémophiles Hôpital Universitaire Purpan, Toulouse
- Germany (7):
  - Charité Campus Virchow Klinikum, Klinik für Pädiatrie m.S. Onkologie und Hämatologie, Berlin
  - Department of Internal Medicine, Hemophilia Treatment Center, Vivantes Klinikum im Friedrichshain, Berlin
  - Institut für Experimentelle Hämatologie und Transfusionsmedizin Universitätsklinikum Bonn, Bonn
  - Klinik Bremen-Mitte Prof.-Hess-Kinderklinik, Bremen
  - Hämophilie Zentrum Rhein Main, Frankfurt
  - University Hospital Frankfurt & Goethe University - Clinical and Molecular Hemostasis, Department of Pediatrics, Frankfurt am Main
  - Dr. v. Haunersches Kinderspital University of Munich, Munich
- Haemophilia-Haemostasis Unit St. Sophia Children's Hospital, Athens, Greece
- Children's Health Ireland (CHI) at Crumlin, Dublin, Ireland
- The National Hemophilia Center Sheba Medical Center, Tel Hashomer, Ramat Gan, Israel
- Italy (3):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Gaslini Hospital, Genova
  - A. Bianchi Bonomi Hemophilia and Thrombosis Centre IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
- Van Creveld Kliniek University Medical Center Utrecht, Utrecht, Netherlands
- Oslo University Hospital, Oslo, Norway
- Centro Hospitalar São João, S. Imuno-hemoterapia, Porto, Portugal
- Spain (4):
  - Unitat Hemofilia Hospital Vall d'Hebron, Barcelona
  - Unidad de Coagulopatías Hospital Universitario La Paz, Madrid
  - Hospital General Unidad de Hemofilia 1 Sur Hospitales Universitarios Virgen del Rocio, Seville
  - Unidad de Coagulopatias Congenitas Hospital Universitario la Fe, Valencia
- Sweden (2):
  - Lund University Hospital, Malmo
  - Department of Pediatrics, Clinic of Coag. Disorders Karolinska Hospital, Stockholm
- Inselspital Bern, University Children's Hospital, Bern, Switzerland
- United Kingdom (4):
  - Birmingham Children's Hospital NHS Trust - Department of Haematology, Birmingham
  - Royal Hospital for Sick Children, Edinburgh
  - Department of Haematology Royal Hospital for Sick Children, Glasgow
  - Haemophila Center Great Ormond Street Hospital for Children, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Kovel M, van Haaster AC, Carcao M, Ranta S, Glosli H, Rivard GE, Kenet G, Kurnik K, Van Geet C, Carvalho M, Andersson NG, Kartal-Kaess M, Ljung R, van den Berg HM; PedNet Study Group. Blood Group O Does Not Increase the Risk of Inhibitors in Severe Haemophilia A: Data from the PedNet Study Group. Haemophilia. 2025 May;31(3):419-423. doi: 10.1111/hae.70035. Epub 2025 Mar 23. PMID 40123267
- [Background] Carcao M, Konigs C, Andersson NG, de Kovel M, de Boer-Verdonk E, Motwani J, Blatny J, Olivieri M, van den Berg M, Fischer K. Predictors of immune tolerance induction success in 231 children with severe hemophilia A with high-titer inhibitors - lessons learned from the PedNet prospective cohort study. J Thromb Haemost. 2025 Oct;23(10):3134-3147. doi: 10.1016/j.jtha.2025.07.010. Epub 2025 Jul 22. PMID 40706963
- [Background] Mendoza A, Rivas I, Hidalgo OB, Cid AR, Olivieri M, Ranta S, Labarque V, Andersson NG, de Kovel M, Alvarez-Roman MT. Impact of Family History of Haemophilia on Diagnosis, Management and Outcomes in Severe Haemophilia. Haemophilia. 2025 Jul;31(4):679-686. doi: 10.1111/hae.70018. Epub 2025 May 30. PMID 40444652
- [Background] Ranta S, Zapotocka E, Andersson NG, Fischer K, Kenet G, de Kovel M, Konigs C, Labarque V, Male C, Olivieri M, Motwani J. A survey on clinical practice in monitoring and management of bleeding in children with haemophilia A on emicizumab prophylaxis in the PedNet centres. Thromb Res. 2025 May;249:109307. doi: 10.1016/j.thromres.2025.109307. Epub 2025 Mar 19. No abstract available. PMID 40120320
- [Background] van den Berg HM, Gouw SC, van der Bom JG. Factor VIII products and inhibitors in severe hemophilia A. N Engl J Med. 2013 Apr 11;368(15):1457. doi: 10.1056/NEJMc1301995. No abstract available. PMID 23574131
- [Background] Gouw SC, van den Berg HM, Fischer K, Auerswald G, Carcao M, Chalmers E, Chambost H, Kurnik K, Liesner R, Petrini P, Platokouki H, Altisent C, Oldenburg J, Nolan B, Garrido RP, Mancuso ME, Rafowicz A, Williams M, Clausen N, Middelburg RA, Ljung R, van der Bom JG; PedNet and Research of Determinants of INhibitor development (RODIN) Study Group. Intensity of factor VIII treatment and inhibitor development in children with severe hemophilia A: the RODIN study. Blood. 2013 May 16;121(20):4046-55. doi: 10.1182/blood-2012-09-457036. Epub 2013 Apr 3. PMID 23553768
- [Background] Carcao MD, van den Berg HM, Ljung R, Mancuso ME; PedNet and the Rodin Study Group. Correlation between phenotype and genotype in a large unselected cohort of children with severe hemophilia A. Blood. 2013 May 9;121(19):3946-52, S1. doi: 10.1182/blood-2012-11-469403. Epub 2013 Mar 12. PMID 23482934
- [Background] Clausen N, Petrini P, Claeyssens-Donadel S, Gouw SC, Liesner R; PedNet and Research of Determinants of Inhibitor development (RODIN) Study Group. Similar bleeding phenotype in young children with haemophilia A or B: a cohort study. Haemophilia. 2014 Nov;20(6):747-55. doi: 10.1111/hae.12470. Epub 2014 Jun 3. PMID 24893572
- [Background] Fischer K, Ljung R, Platokouki H, Liesner R, Claeyssens S, Smink E, van den Berg HM. Prospective observational cohort studies for studying rare diseases: the European PedNet Haemophilia Registry. Haemophilia. 2014 Jul;20(4):e280-6. doi: 10.1111/hae.12448. Epub 2014 May 2. PMID 24784937
- [Background] Gouw SC, van der Bom JG, Ljung R, Escuriola C, Cid AR, Claeyssens-Donadel S, van Geet C, Kenet G, Makipernaa A, Molinari AC, Muntean W, Kobelt R, Rivard G, Santagostino E, Thomas A, van den Berg HM; PedNet and RODIN Study Group. Factor VIII products and inhibitor development in severe hemophilia A. N Engl J Med. 2013 Jan 17;368(3):231-9. doi: 10.1056/NEJMoa1208024. PMID 23323899
- [Background] Andersson NG, Auerswald G, Barnes C, Carcao M, Dunn AL, Fijnvandraat K, Hoffmann M, Kavakli K, Kenet G, Kobelt R, Kurnik K, Liesner R, Makipernaa A, Manco-Johnson MJ, Mancuso ME, Molinari AC, Nolan B, Perez Garrido R, Petrini P, Platokouki HE, Shapiro AD, Wu R, Ljung R. Intracranial haemorrhage in children and adolescents with severe haemophilia A or B - the impact of prophylactic treatment. Br J Haematol. 2017 Oct;179(2):298-307. doi: 10.1111/bjh.14844. Epub 2017 Jul 12. PMID 28699675
- [Background] Mancuso ME, Fischer K, Santagostino E, Oldenburg J, Platokouki H, Konigs C, Escuriola-Ettingshausen C, Rivard GE, Cid AR, Carcao M, Ljung R, Petrini P, Altisent C, Kenet G, Liesner R, Kurnik K, Auerswald G, Chambost H, Makipernaa A, Molinari AC, Williams M, van den Berg HM; European Pediatric Network for Haemophilia Management (PedNet) the REMAIN (REal life MAnagement of children with INhibitors) Study Group. Risk Factors for the Progression from Low to High Titres in 260 Children with Severe Haemophilia A and Newly Developed Inhibitors. Thromb Haemost. 2017 Dec;117(12):2274-2282. doi: 10.1160/TH17-01-0059. Epub 2017 Dec 6. PMID 29212115
- [Background] Andersson NG, Chalmers EA, Kenet G, Ljung R, Makipernaa A, Chambost H; PedNet Haemophilia Research Foundation. Mode of delivery in hemophilia: vaginal delivery and Cesarean section carry similar risks for intracranial hemorrhages and other major bleeds. Haematologica. 2019 Oct;104(10):2100-2106. doi: 10.3324/haematol.2018.209619. Epub 2019 Feb 21. PMID 30792204
- [Background] van den Berg HM, Fischer K, Carcao M, Chambost H, Kenet G, Kurnik K, Konigs C, Male C, Santagostino E, Ljung R; PedNet Study Group. Timing of inhibitor development in more than 1000 previously untreated patients with severe hemophilia A. Blood. 2019 Jul 18;134(3):317-320. doi: 10.1182/blood.2019000658. Epub 2019 Jun 11. No abstract available. PMID 31186271
- [Background] Male C, Andersson NG, Rafowicz A, Liesner R, Kurnik K, Fischer K, Platokouki H, Santagostino E, Chambost H, Nolan B, Konigs C, Kenet G, Ljung R, Van den Berg M. Inhibitor incidence in an unselected cohort of previously untreated patients with severe haemophilia B: a PedNet study. Haematologica. 2021 Jan 1;106(1):123-129. doi: 10.3324/haematol.2019.239160. PMID 31919092
- [Background] van den Berg HM, Mancuso ME, Konigs C, D'Oiron R, Platokouki H, Mikkelsen TS, Motwani J, Nolan B, Santagostino E; European Pediatric Network for Haemophilia Management (PedNet). ITI Treatment is not First-Choice Treatment in Children with Hemophilia A and Low-Responding Inhibitors: Evidence from a PedNet Study. Thromb Haemost. 2020 Aug;120(8):1166-1172. doi: 10.1055/s-0040-1713097. Epub 2020 Jun 22. PMID 32572865
- [Background] Andersson NG, Wu R, Carcao M, Claeyssens-Donadel S, Kobelt R, Liesner R, Makipernaa A, Ranta S, Ljung R; ICH study group. Long-term follow-up of neonatal intracranial haemorrhage in children with severe haemophilia. Br J Haematol. 2020 Jul;190(2):e101-e104. doi: 10.1111/bjh.16740. Epub 2020 Jun 9. No abstract available. PMID 32519345
- [Background] Platokouki H, Fischer K, Gouw SC, Rafowicz A, Carcao M, Kenet G, Liesner R, Kurnik K, Rivard GE, van den Berg HM. Vaccinations are not associated with inhibitor development in boys with severe haemophilia A. Haemophilia. 2018 Mar;24(2):283-290. doi: 10.1111/hae.13387. Epub 2017 Dec 15. PMID 29243367
- [Background] Khair K, Ranta S, Thomas A, Lindvall K; PedNet study group. The impact of clinical practice on the outcome of central venous access devices in children with haemophilia. Haemophilia. 2017 Jul;23(4):e276-e281. doi: 10.1111/hae.13241. Epub 2017 May 24. PMID 28544163
- [Background] Hashemi SM, Fischer K, Moons KGM, van den Berg HM; PedNet Study group. Validation of the prediction model for inhibitor development in PUPs with severe haemophilia A. Haemophilia. 2016 Mar;22(2):e116-e118. doi: 10.1111/hae.12895. Epub 2016 Feb 8. No abstract available. PMID 26856685
- [Background] Ranta S, Motwani J, Blatny J, Buhrlen M, Carcao M, Chambost H, Escuriola C, Fischer K, Kartal-Kaess M, de Kovel M, Kenet G, Male C, Nolan B, d'Oiron R, Olivieri M, Zapotocka E, Andersson NG, Konigs C. Dilemmas on emicizumab in children with haemophilia A: A survey of strategies from PedNet centres. Haemophilia. 2023 Sep;29(5):1291-1298. doi: 10.1111/hae.14847. Epub 2023 Aug 30. PMID 37647211
- [Background] Labarque V, Mancuso ME, Kartal-Kaess M, Ljung R, Mikkelsen TS, Andersson NG. F8/F9 variants in the population-based PedNet Registry cohort compared with locus-specific genetic databases of the European Association for Haemophilia and Allied Disorders and the Centers for Disease Control and Prevention Hemophilia A or Hemophilia B Mutation Project. Res Pract Thromb Haemost. 2023 Jan 10;7(1):100036. doi: 10.1016/j.rpth.2023.100036. eCollection 2023 Jan. PMID 36798899
- [Background] Fischer K, Carcao M, Male C, Ranta S, Pergantou H, Kenet G, Kartal-Kaess M, Konigs C, Carvalho M, Alvarez MT, Brakenhoff T, Chambost H, van den Berg HM. Different inhibitor incidence for individual factor VIII concentrates in 1076 previously untreated patients with severe hemophilia A: data from the PedNet cohort. J Thromb Haemost. 2023 Mar;21(3):700-703. doi: 10.1016/j.jtha.2022.11.020. Epub 2022 Dec 22. No abstract available. PMID 36696215
- [Background] Ljung R, de Kovel M, van den Berg HM; PedNet study group. Primary prophylaxis in children with severe haemophilia A and B-Implementation over the last 20 years as illustrated in real-world data in the PedNet cohorts. Haemophilia. 2023 Mar;29(2):498-504. doi: 10.1111/hae.14729. Epub 2022 Dec 26. PMID 36571801
- [Background] Schmidt DE, Michalopoulou A, Fischer K, Motwani J, Andersson NG, Pergantou H, Ranta S; PedNet Study Group. Long-term joint outcomes in adolescents with moderate or severe haemophilia A. Haemophilia. 2022 Nov;28(6):1054-1061. doi: 10.1111/hae.14636. Epub 2022 Aug 4. PMID 35925557
- [Background] Alvarez-Roman MT, Kurnik K; PedNet Study Group. Care for children with haemophilia during COVID-19: Data of the PedNet study group. Haemophilia. 2021 Jul;27(4):e537-e539. doi: 10.1111/hae.14286. Epub 2021 Mar 8. No abstract available. PMID 33683753
- [Background] Minna K, Anne M, Beatrice N, Rainer K, Susanna R. Correction of haemostasis can be reduced to four days for CVAD implantation in severe haemophilia A patients: Data from the PedNet study group. Haemophilia. 2021 May;27(3):392-397. doi: 10.1111/hae.14231. Epub 2021 Mar 21. PMID 33745218
- [Background] Andersson NG, Labarque V, Letelier A, Mancuso ME, Buhrlen M, Fischer K, Kartal-Kaess M, Koskenvuo M, Mikkelsen T, Ljung R; PedNet study group. Novel F8 and F9 gene variants from the PedNet hemophilia registry classified according to ACMG/AMP guidelines. Hum Mutat. 2020 Dec;41(12):2058-2072. doi: 10.1002/humu.24117. Epub 2020 Oct 14. PMID 32935414
- [Background] Jonker CJ, Oude Rengerink K, Hoes AW, Mol PGM, van den Berg HM. Inhibitor development in previously untreated patients with severe haemophilia: A comparison of included patients and outcomes between a clinical study and a registry-based study. Haemophilia. 2020 Sep;26(5):809-816. doi: 10.1111/hae.14100. Epub 2020 Jul 6. PMID 32627880
- [Background] Andersson NG, Labarque V, Kartal-Kaess M, Pinto F, Mikkelsen TS, Ljung R, Group PS. Factor VIII genotype and the risk of developing high-responding or low-responding inhibitors in severe hemophilia A: data from the PedNet Hemophilia Cohort of 1,202 children. Haematologica. 2024 Apr 1;109(4):1293-1296. doi: 10.3324/haematol.2023.284095. No abstract available. PMID 37881836
- [Background] Fischer K, Kenet G, Kurnik K, Carcao M, Oldenburg J, Stamm-Mikkelsen T, Cid Haro AR, Koskenvuo M, Blatny J, Konigs C. Determinants of bleeding before and during immune tolerance in 222 boys with severe hemophilia A and inhibitors >5 BU. Blood Adv. 2024 Jan 23;8(2):369-377. doi: 10.1182/bloodadvances.2023011442. PMID 38214949
- [Background] van der Zwet K, de Kovel M, Motwani J, van Geet C, Nolan B, Glosli H, Escuriola Ettingshausen C, Konigs C, Kenet G, Fischer K; PedNet Investigators. Bleeding control improves after switching to emicizumab: Real-world experience of 177 children in the PedNet registry. Haemophilia. 2024 May;30(3):685-692. doi: 10.1111/hae.15015. Epub 2024 Apr 5. PMID 38578720
- [Background] de Kovel MS, Escuriola-Ettingshausen C, Konigs C, Ranta S, Fischer K; PedNet Study Group. Bleeding phenotype according to factor level in 825 children with nonsevere hemophilia: data from the PedNet cohort. J Thromb Haemost. 2024 Sep;22(9):2460-2469. doi: 10.1016/j.jtha.2024.05.030. Epub 2024 Jun 10. PMID 38866249
- See also: Website of the PedNet Registry — http://www.pednet.eu